CLINICAL TRIAL: NCT06689007
Title: Stimulating Change in Pediatric Rehabilitation: An Implementation Intervention to Increase Use of Functional Electrical Stimulation
Brief Title: FES Implementation Pediatrics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Kristin Musselman, Associate Professor, University of Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 46640
Record Dates: First submitted 2024-11-12; First posted 2024-11-14 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Cerebral Palsy (CP)
Keywords: functional electrical stimulation; implementation intervention; physical therapist; occupational therapist
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Implementation Intervention (Experimental)
  Interventions: Other: Implementation Intervention

INTERVENTIONS:
Other: Implementation Intervention — The intervention employs four established implementation strategies according to the Expert Recommendations for Implementing Change: conduct educational meetings, provide ongoing consultation, provide technical assistance, and change physical structure and equipment. The first component is a six-week online course led by the PI that combines weekly pre-recorded lectures, hands-on activities, group mentoring sessions and a reflective assignment. The second component of the intervention is ensuring access to the equipment needed for FES. The third component of the intervention is access to the FES Toolkit.

SUMMARY:
Physical rehabilitation interventions that promote activity-dependent neuroplasticity are desired for children with CP as this will result in improved motor skill and function. In adult neurological populations, such as stroke and spinal cord injury, FES is a recommended, evidence-based intervention that addresses motor and sensory impairments and promotes neuroplasticity. The evidence base supporting the safety, feasibility and efficacy of FES for youth with CP is rapidly growing, yet FES is not commonly used in Canadian pediatric rehabilitation. Through interviews with Canadian pediatric physical and occupational therapists, we identified numerous barriers to FES implementation, including a lack of knowledge and training in FES, difficulty accessing FES equipment, and a perceived lack of time to deliver FES within a treatment session. To address these barriers, we have developed an implementation intervention for FES that consists of an online course and toolkit for physical and occupational therapists. As a next step, we will evaluate the effects of the implementation intervention on pediatric therapists' knowledge, confidence and use of FES.

ELIGIBILITY:
Inclusion Criteria:

1. Licensed to practice physical or occupational therapy in Canada.
2. Report that CP comprises ≥20% of their caseload over the past year.
3. Has not previously taken a continuing education course in FES.
4. Reports never (0% of treatment sessions) or rarely (1-20% of treatment sessions) using neuromuscular electrical stimulation (NMES) or FES in their clinical practice.
5. Report being able to participate in a six-week online FES course from October 18 2024 - November 28 2024.
6. Able to complete the course and interview in English.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-07-18 (Actual); Study Completion 2025-07-18 (Actual)

PRIMARY OUTCOMES:
FES knowledge quiz | From pre-intervention to immediately post-intervention and six months post-intervention
FES Confidence Questionnaire | From pre-intervention to immediately post-intervention and six months post-intervention
FES Use Survey | From pre-intervention to immediately post-intervention and six months post-intervention
Technology Assistance Model 2 Questionnaire | From pre-intervention to immediately post-intervention and six months post-intervention
Semi-structured Interview | Six months post-intervention
  Guided by the RE-AIM Framework

CONTACTS AND LOCATIONS:
Locations (1):
- University of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided